CLINICAL TRIAL: NCT04033367
Title: A Randomized Double-blind, Placebo-controlled Study Evaluating the Effect of Dupilumab on Sleep in Adult Patients With Moderate to Severe Atopic Dermatitis (AD)
Brief Title: SAR231893-LPS15497- "Dupilumab Effect on Sleep in AD Patients"
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LPS15497; 2018-004705-26 (EudraCT Number); U1111-1223-4147 (Other: UTN)
Record Dates: First submitted 2019-07-16; First posted 2019-07-26 (Actual); Results first posted 2022-11-02 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dupilumab/Dupilumab (Experimental): Participants received dupilumab 600 milligrams (mg) (loading dose) injection subcutaneously (SC) on Day 1 followed by dupilumab 300 mg injection SC every 2 weeks (q2w) up to Week 10 in the double-blind (DB) period of 12 weeks. After completion of DB period, participants entered in the open-label extension (OLE) period (Week 12 to 24) and continued to receive dupilumab 300 mg injection SC q2w from Week 12 up to Week 22.
  Interventions: Drug: Dupilumab
- Placebo/Dupilumab (Placebo Comparator): Participants received placebo matching to dupilumab injection SC on Day 1 then followed by placebo injection SC q2w up to Week 10 in the DB period of 12 weeks. After completion of DB period, participants entered in the OLE period (Week 12 to 24) and received dupilumab 600 mg (loading dose) at Week 12 followed by dupilumab 300 mg injection SC q2w up to Week 22.
  Interventions: Drug: Dupilumab; Drug: Placebo

INTERVENTIONS:
Drug: Dupilumab — Pharmaceutical form: solution for injection Route of administration: subcutaneous
  Other Names: SAR231893
Drug: Placebo — Pharmaceutical form: solution for injection Route of administration: subcutaneous
  Arms: Placebo/Dupilumab

SUMMARY:
Primary Objective:

To evaluate the effect of dupilumab on sleep quality in adult participants with moderate to severe atopic dermatitis (AD).

Secondary Objectives:

To evaluate the effect of dupilumab on objective and subjective quantitative sleep parameters, AD related outcomes, and daytime consequences of sleep deprivation.

To continue to assess the safety and tolerability throughout the study.

DETAILED DESCRIPTION:
Duration per participant was up to 28 weeks.

ELIGIBILITY:
Inclusion criteria:

Participants, male or female 18 years or older,

* with diagnosed chronic AD, demonstrated 1) inadequate response to topical medications, 2) expected severity of AD and 3) sleep disturbance.
* had applied skin emollients (moisturizers) at least 7 days before screening.
* had applied medium potency topical corticosteroids (TCS) on all active AD lesions at least 7 days before screening.
* willed and able to comply with all clinic visits and study-related procedures.
* provided signed informed consent.

Exclusion criteria:

Participants excluded from the study:

* with known hypersensitivity to Dupixent, clinical depression, drug abuse history, sleep problems not related to AD, irregular sleep pattern, active/acute infections, severe medical conditions, laboratory abnormalities, any condition that might present unreasonable risk to participants or interfered with study assessment, or any severe concomitant illness(es) that would adversely affect the participant's participation in the study, and contraindications of topical corticosteroids.
* at Baseline, presence of any conditions listed as criteria for study drug discontinuation.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (42):
- United States (8):
  - Investigational Site Number :8400012, North Little Rock, Arkansas
  - Investigational Site Number :8400002, Redwood City, California
  - Investigational Site Number :8400001, Rolling Hills Estates, California
  - Investigational Site Number :8400013, Colorado Springs, Colorado
  - Investigational Site Number :8400005, Denver, Colorado
  - Investigational Site Number :8400003, Sarasota, Florida
  - Investigational Site Number :8400007, Medford, Oregon
  - Investigational Site Number :8400008, Charleston, South Carolina
- Australia (4):
  - Investigational Site Number :0360006, Phillip, Australian Capital Territory
  - Investigational Site Number :0360001, Kogarah, New South Wales
  - Investigational Site Number :0360007, Woolloongabba, Queensland
  - Investigational Site Number :0360003, Carlton, Victoria
- France (4):
  - Investigational Site Number :2500001, Brest
  - Investigational Site Number :2500003, Nantes
  - Investigational Site Number :2500002, Paris
  - Investigational Site Number :2500006, Toulouse
- Germany (5):
  - Investigational Site Number :2760005, Bad Bentheim
  - Investigational Site Number :2760002, Frankfurt am Main
  - Investigational Site Number :2760006, Friedrichshafen
  - Investigational Site Number :2760001, Göttingen
  - Investigational Site Number :2760004, Münster
- Israel (2):
  - Investigational Site Number :3760005, Afula
  - Investigational Site Number :3760003, Jerusalem
- Italy (6):
  - Investigational Site Number :3800005, Rozzano, Milano
  - Investigational Site Number :3800006, Perugia
  - Investigational Site Number :3800001, Pisa
  - Investigational Site Number :3800004, Reggio Calabria
  - Investigational Site Number :3800002, Roma
  - Investigational Site Number :3800003, Siena
- Spain (8):
  - Investigational Site Number :7240004, Granada, Andalusia
  - Investigational Site Number :7240001, Barcelona / Sabadell, Castille and León
  - Investigational Site Number :7240003, Manises, Valencia
  - Investigational Site Number :7240006, Córdoba
  - Investigational Site Number :7240008, Madrid
  - Investigational Site Number :7240010, Madrid
  - Investigational Site Number :7240005, Seville
  - Investigational Site Number :7240002, Valencia
- Investigational Site Number :7560001, Bern, Switzerland
- United Arab Emirates (2):
  - Investigational Site Number :7840002, Abu Dhabi
  - Investigational Site Number :7840001, Dubai
- United Kingdom (2):
  - Investigational Site Number :8260002, Dudley, Birmingham
  - Investigational Site Number :8260004, Edinburgh, Edinburgh, City of

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LPS15497 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25275&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 46 centers in 10 countries. A total of 267 participants were screened between 22 August 2019 and 13 April 2021, of which 188 participants were enrolled and randomized. A total of 79 participants failed screening mainly due to not meeting eligibility criteria.
Pre-assignment Details: Participants were randomly assigned to receive either dupilumab or placebo in a 2:1 ratio via interactive voice response system.
Period: DB Period (Up to Week 12)
Arm/Group | Dupilumab/Dupilumab | Placebo/Dupilumab
Started | 127 | 61
Completed | 122 | 60
Not Completed | 5 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 4 | 0
Period: OLE Period (Week 12 to Week 24)
Arm/Group | Dupilumab/Dupilumab | Placebo/Dupilumab
Started | 122 | 60
Completed | 117 | 59
Not Completed | 5 | 1
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Other-unspecified | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on intent-to-treat (ITT) analysis set which included all randomized participants with a treatment kit number allocated and recorded in the interactive response technology (IRT) database, regardless of whether the treatment kit was used or not and were analyzed according to the treatment group allocated by randomization.
Groups:
- Dupilumab/Dupilumab: Participants received dupilumab 600 mg (loading dose) injection SC on Day 1 followed by dupilumab 300 mg injection SC q2w up to Week 10 in the DB period of 12 weeks. After completion of DB period, participants entered in the OLE period (Week 12 to 24) and continued to receive dupilumab 300 mg injection SC q2w from Week 12 up to Week 22.
- Total: Total of all reporting groups
Arm/Group | Dupilumab/Dupilumab | Placebo/Dupilumab | Total
Number analyzed (Participants) | 127 | 61 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (14.68) | 34.5 (15.36) | 35.7 (14.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 31 | 97
  Male | 61 | 30 | 91
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 11 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 1 | 7
  White | 103 | 46 | 149
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: DB Period: Percent Change From Baseline in Sleep Quality Numerical Rating Scale (NRS) at Week 12
Description: Sleep quality NRS was used to assess the quality of the participant's previous night's sleep. It was collected on a 11-point scale ranged from 0 (worst possible sleep) to 10 (best possible sleep), where higher score indicated better outcome. Percent change from Baseline in sleep quality NRS at Week 12 was reported in this outcome measure.
Time Frame: Baseline, Week 12
Population: Analysis was performed on modified intent-to-treat (mITT) analysis set which included all randomized participants with a treatment kit number allocated and recorded in the IRT database, regardless of whether the treatment kit was used or not, who had a Baseline and at least one post-baseline measurement. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- DB Period: Dupilumab: Participants received dupilumab 600 mg (loading dose) injection SC on Day 1 followed by dupilumab 300 mg injection SC q2w up to Week 10.
- DB Period: Placebo: Participants received placebo matching to dupilumab injection SC on day 1 then followed by placebo injection SC q2w up to Week 10.
Arm/Group | DB Period: Dupilumab | DB Period: Placebo
Number analyzed (Participants) | 122 | 60
percent change | -47.71 (27.240) | -32.98 (29.536)
Statistical Analysis 1: Comparison: DB Period: Dupilumab vs DB Period: Placebo; A hierarchical testing procedure was used to control the overall type I error. Testing was then performed sequentially in order the outcome measures are reported and continued when primary outcome measure was statistically significant at two-sided 0.05 level; Test type: Superiority; p < 0.001, Mixed Models Analysis — Threshold of significance at 0.05; Least square mean difference = -15.52, 95% CI 2-sided [-24.13 to -6.90] — Dupilumab versus Placebo

2. Secondary Outcome: DB Period: Percent Change From Baseline in Peak Pruritus NRS at Week 12
Description: Peak Pruritus NRS was an assessment tool that was used by participants to report the intensity of their pruritus (itch) during a 24-hour recall period. Participants were asked the following question: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?". Participants answered the question at the specified time point (for the last 24 hours) on the scale of 0 (no itch) to 10 (worst itch imaginable), where higher scores indicated greater severity.
Time Frame: Baseline, Week 12
Population: Analysis was performed on mITT set. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | DB Period: Dupilumab | DB Period: Placebo
Number analyzed (Participants) | 110 | 48
percent change | -52.45 (30.614) | -23.29 (30.075)
Statistical Analysis 1: Comparison: DB Period: Dupilumab vs DB Period: Placebo; A hierarchical testing procedure was used to control the overall type I error. Testing was then performed sequentially in order the outcome measures are reported and continued when previous outcome measure was statistically significant at two-sided 0.05 level; Test type: Superiority; p < 0.001, Mixed Models Analysis — Threshold of significance at 0.05; Least square mean difference = -27.87, 95% CI 2-sided [-37.96 to -17.78] — Dupilumab versus Placebo

3. Secondary Outcome: DB Period: Change From Baseline in SCORing Atopic Dermatitis (SCORAD) Total Score at Week 12
Description: SCORAD is a validated scoring index for AD, which consists of 3 components i.e., A =extent or affected body surface area (BSA) assessed as a percentage of each defined body area and reported as the sum of all areas, with a maximum score of 100%. B=severity of 6 specific symptoms of AD (redness, swelling, oozing/crusting, excoriation, skin thickening/lichenification, dryness) assessed using the following scale: none (0), mild (1), moderate (2), or severe (3) (for a maximum of 18 total points) and C=subjective symptoms scored by participants on VAS, where "0" is no itch (or no sleeplessness) and "10" is the worst imaginable itch (or sleeplessness) with a maximum score of 20. SCORAD total score was calculated using these 3 aspects: extent (A: 0-100), severity (B: 0-18), and subjective symptoms (C: 0-20) using the formula: A/5 + 7*B/2+ C to give the SCORAD total score range of 0 to 103, where 0 = no disease to 103 = severe disease. Higher values of SCORAD represent worse outcome.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DB Period: Dupilumab | DB Period: Placebo
Number analyzed (Participants) | 109 | 48
score on a scale | -37.78 (17.743) | -20.55 (17.944)
Statistical Analysis 1: Comparison: DB Period: Dupilumab vs DB Period: Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis — Threshold of significance at 0.05; Least square mean difference = -15.06, 95% CI 2-sided [-20.56 to -9.56] — Dupilumab versus Placebo

4. Secondary Outcome: DB Period: Change From Baseline in SCORAD Sleep Loss Visual Analog Scale (VAS) Score at Week 12
Description: SCORAD is a validated scoring index for AD, which combines extent (A, 0-100), severity (B, 0-18), and subjective symptoms (C, 0-20) based on itch and sleeplessness, each scored (0-10). The SCORAD for an individual was calculated by the formula: A/5 + 7B/2 + C (can range from 0 to 103). Subjective symptoms (i.e., itch and sleeplessness/sleep loss) were each scored by the participant using a VAS ranging from 0 to 10, where "0" is no itch (or no sleep loss) and "10" is the worst imaginable itch (or sleeplessness). Change from Baseline in SCORAD sleeplessness/sleep loss VAS score is reported in this outcome measure.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DB Period: Dupilumab | DB Period: Placebo
Number analyzed (Participants) | 108 | 47
score on a scale | -4.85 (2.953) | -2.31 (3.024)
Statistical Analysis 1: Comparison: DB Period: Dupilumab vs DB Period: Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis — Threshold of significance at 0.05; Least square mean difference = -2.08, 95% CI 2-sided [-2.97 to -1.18] — Dupilumab versus Placebo

5. Secondary Outcome: DB Period: Change From Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Related Impairment Short Form 8a (SF8a) Total T-Score at Week 12
Description: PROMIS is a Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), Level 2, sleep disturbance measure. In this study, 8- item PROMIS Sleep Related Impairment SF8a that assesses the domain of sleep related impairment in the past 7 days in individuals aged 18 and older, was used. Each item asks the participant to rate the severity of the participant's sleep related impairment during the past 7 days (at each specified visit) on a 5-point scale (1 = not at all; 2 = a little bit; 3 = somewhat; 4 = quite a bit; and 5 = very much) with raw score ranging from 8 to 40; higher scores indicating greater severity of sleep impairment. PROMIS T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation of 10. Possible range for T-score is 30 to 80, with higher scores indicating greater severity of sleep impairment.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | DB Period: Dupilumab | DB Period: Placebo
Number analyzed (Participants) | 103 | 54
T-score | -11.42 (6.710) | -7.77 (7.240)
Statistical Analysis 1: Comparison: DB Period: Dupilumab vs DB Period: Placebo; A hierarchical testing procedure was used to control the overall type I error. Testing was then performed sequentially in order the outcome measures are reported and continued when previous outcome measure was statistically significant at two-sided 0.05; Test type: Superiority; p < 0.001, Mixed Models Analysis — Threshold of significance at 0.05; Least square mean difference = -3.61, 95% CI 2-sided [-5.68 to -1.53] — Dupilumab versus Placebo

6. Secondary Outcome: DB Period: Change From Baseline in Weekly Average Total Sleep Time (TST) at Week 12
Description: A sleep diary was designed to gather information about participant's daily sleep pattern. It measured night-time sleep assessments. TST (in minutes) was calculated using the formula: Time of waking up for the day minus time of falling sleep minus Wake After Sleep Onset (WASO), where WASO = time awake after initial sleep onset but before the final awakening for the day. Data for WASO was collected from Question 3 of the Sleep Diary: "Considering all the times you woke up last night, how much time were you awake in total?". Baseline and Post-baseline weekly average data were calculated based on the mean of the data over the 7 days prior to and including the day at the Baseline or at the end of the corresponding week. In this outcome measure, change from Baseline in TST at Week 12 is reported.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | DB Period: Dupilumab | DB Period: Placebo
Number analyzed (Participants) | 108 | 47
minutes | 9.00 (70.987) | -6.36 (55.620)
Statistical Analysis 1: Comparison: DB Period: Dupilumab vs DB Period: Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.297, Mixed Models Analysis — Threshold of significance at 0.05; Least square mean difference = 9.97, 95% CI 2-sided [-8.86 to 28.79] — Dupilumab versus Placebo

7. Secondary Outcome: DB Period: Change From Baseline in Weekly Average Sleep Efficiency (SE) at Week 12
Description: A sleep diary was designed to gather information about participant's daily sleep pattern. It measured night-time sleep assessments. SE was calculated using the formula: (TST divided by [Time of waking up for the day - Time of trying to fall sleep]) multiplied by 100 percent (%). TST (in minutes) was calculated using the formula: Time of waking up for the day minus time of falling sleep minus Wake After Sleep Onset (WASO), where WASO = time awake after initial sleep onset but before the final awakening for the day. Baseline and Post-baseline weekly average data were calculated based on the mean of the data over the 7 days prior to and including the day at the Baseline or at the end of the corresponding week. In this outcome measure, change from Baseline in SE at Week 12 is reported.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of time in bed spent asleep
Arm/Group | DB Period: Dupilumab | DB Period: Placebo
Number analyzed (Participants) | 108 | 47
percentage of time in bed spent asleep | 1.81 (6.593) | 1.53 (6.018)

8. Secondary Outcome: DB Period: Change From Baseline in Weekly Average Wake After Sleep Onset (WASO) at Week 12
Description: A sleep diary was designed to gather information about participant's daily sleep pattern. It measured night-time sleep assessments. WASO = time awake (in minutes) after initial sleep onset but before the final awakening for the day. Data for WASO was collected from Question 3 of the Sleep Diary: "Considering all the times you woke up last night, how much time were you awake in total?". Baseline and Post-baseline weekly average data were calculated based on the mean of the data over the 7 days prior to and including the day at the Baseline or at the end of the corresponding week. In this outcome measure, change from Baseline in WASO at Week 12 is reported.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | DB Period: Dupilumab | DB Period: Placebo
Number analyzed (Participants) | 108 | 47
minutes | -6.79 (22.786) | -9.19 (24.661)

9. Secondary Outcome: DB Period: Change From Baseline in Weekly Average Sleep Onset Latency (SOL) at Week 12
Description: A sleep diary was designed to gather information about participant's daily sleep pattern. It measured night-time sleep assessments. SOL (in minutes) was calculated using the formula: Time of falling sleep - Time of trying to fall sleep. Baseline and Post-baseline weekly average data were calculated based on the mean of the data over the 7 days prior to and including the day at the Baseline or at the end of the corresponding week. In this outcome measure, change from Baseline in SOL at Week 12 is reported.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | DB Period: Dupilumab | DB Period: Placebo
Number analyzed (Participants) | 108 | 47
minutes | -1.44 (19.983) | -3.37 (21.477)

10. Secondary Outcome: DB Period: Percentage of Participants With Eczema Area Severity Index-50 (EASI-50) (Greater Than or Equal to [>=] 50% Improvement From Baseline) at Week 12
Description: EASI evaluates severity of participants with AD (excluded scalp, palms, soles) based on severity of AD clinical signs and % of body surface area (BSA) affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin] and lower limbs [including buttocks]) on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % BSA with AD in each body region: 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), and 6 (90% to 100%). Total EASI score ranged from 0.0 to 72.0, higher scores = greater severity of AD. Percentage of participants with EASI-50 (>=50% improvement from Baseline in EASI score) at Week 12 is reported in this outcome measure.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | DB Period: Dupilumab | DB Period: Placebo
Number analyzed (Participants) | 109 | 48
percentage of participants | 89.0 | 58.3

11. Secondary Outcome: DB Period: Percentage of Participants With Eczema Area Severity Index-75 (EASI-75) (>= 75% Improvement From Baseline) at Week 12
Description: EASI evaluates severity of participants with AD (excluded scalp, palms, soles) based on severity of AD clinical signs and % BSA affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin] and lower limbs [including buttocks]) on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % BSA with AD in each body region: 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), and 6 (90% to 100%). Total EASI score ranged from 0.0 to 72.0, higher scores = greater severity of AD. Percentage of participants with EASI-75 (>=75% improvement from Baseline in EASI score) at Week 12 is reported in this outcome measure.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | DB Period: Dupilumab | DB Period: Placebo
Number analyzed (Participants) | 109 | 48
percentage of participants | 60.6 | 29.2

12. Secondary Outcome: DB Period: Change From Baseline in Patient Oriented Eczema Measure (POEM) Total Score at Week 12
Description: The POEM was a 7-item, validated questionnaire used in clinical practice and clinical trials to assess disease symptoms in children and adults with AD. The format is participant response to 7 items (dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping) based on symptom frequency during the past week (i.e., 0 = 'no days', 1 = '1 to 2 days', 2 = '3 to 4 days', 3 = '5 to 6' days, and 4 = 'every day'). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (severe disease). Higher scores indicated more severe disease and poor quality of life.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DB Period: Dupilumab | DB Period: Placebo
Number analyzed (Participants) | 90 | 39
score on a scale | -13.63 (7.496) | -4.44 (6.824)

13. Secondary Outcome: DB Period: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score at Week 12
Description: DLQI was a 10-item questionnaire that measures the impact of skin disease. Each question was evaluated on a 4-point scale ranged from 0 to 3 where, 0 = not at all, 1= a little, 2= a lot, 3= very much, where higher scores indicated more impact on quality of life. Scores from all 10 questions were added up to give DLQI total score range from 0 (not at all) to 30 (very much). Higher scores indicated more impact on quality of life of participants.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DB Period: Dupilumab | DB Period: Placebo
Number analyzed (Participants) | 90 | 39
score on a scale | -11.82 (6.503) | -7.54 (6.801)

14. Secondary Outcome: DB Period: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily have to have a causal relationship with the treatment. Serious adverse events (SAEs) were defined as any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were defined as AEs that developed, worsened or became serious during the TEAE period (from the first investigational medicinal product [IMP] administration to the last IMP administration + 14 days) in DB period.
Time Frame: Baseline up to 14 days after last IMP administration (i.e., up to Week 12)
Population: Analysis was performed on safety analysis set (SAS) which included all randomized participants who actually received at least 1 dose or partial dose of the IMP and analyzed according to the treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Dupilumab | DB Period: Placebo
Number analyzed (Participants) | 127 | 61
Participants
  Any TEAEs | 72 | 41
  Any TESAEs | 2 | 1

15. Secondary Outcome: Entire Study Duration: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily have to have a causal relationship with the treatment. SAEs were defined as any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were defined as AEs that developed, worsened or became serious during the TEAE period (from the first IMP administration to the last IMP administration + 14 days).
Time Frame: Baseline up to 14 days after last IMP administration (i.e., up to Week 24)
Population: Analysis was performed on SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Dupilumab/Dupilumab | Placebo/Dupilumab
Number analyzed (Participants) | 127 | 61
Participants
  Any TEAEs | 89 | 46
  Any TESAEs | 3 | 1

ADVERSE EVENTS:
Time Frame: From the first IMP administration up to Week 12 (for DB period arms) and from first IMP administration in OLE period up to Week 24 (for OLE period arms)
Description: Reported AEs were TEAEs that occurred/worsened in grade or became serious during TEAE period (defined as the time from the first IMP administration in DB period to the last IMP administration in OLE period + 14 days). Analysis was performed on SAS.
Groups:
- OLE Period: Placebo/Dupilumab: Participants received placebo matching to dupilumab injection SC on Day 1 then followed by placebo injection SC q2w up to Week 10 in the DB period of 12 weeks. After completion of DB period, participants entered in the OLE period (Week 12 to 24) and received dupilumab 600 mg (loading dose) at Week 12 followed by dupilumab 300 mg injection SC q2w up to Week 22.
- OLE Period: Dupilumab/Dupilumab: Participants received dupilumab 600 mg (loading dose) injection SC on Day 1 followed by dupilumab 300 mg injection SC q2w up to Week 10 in the DB period of 12 weeks. After completion of DB period, participants entered in the OLE period (Week 12 to 24) and continued to receive dupilumab 300 mg injection SC q2w from Week 12 up to Week 22.
Arm/Group | DB Period: Placebo | DB Period: Dupilumab | OLE Period: Placebo/Dupilumab | OLE Period: Dupilumab/Dupilumab
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/127 | 0/60 | 0/122
Serious Adverse Events (participants affected / at risk) | 1/61 | 2/127 | 0/60 | 1/122
Other Adverse Events (participants affected / at risk) | 18/61 | 26/127 | 17/60 | 24/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB Period: Placebo (N=61) | DB Period: Dupilumab (N=127) | OLE Period: Placebo/Dupilumab (N=60) | OLE Period: Dupilumab/Dupilumab (N=122)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple Fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB Period: Placebo (N=61) | DB Period: Dupilumab (N=127) | OLE Period: Placebo/Dupilumab (N=60) | OLE Period: Dupilumab/Dupilumab (N=122)
Conjunctivitis (Infections and infestations) | 3 (3) | 12 (12) | 7 (7) | 3 (3)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2) | 4 (4) | 2 (2)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 6 (6) | 15 (15)
Headache (Nervous system disorders) | 5 (5) | 9 (10) | 3 (3) | 2 (2)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 8 (10) | 4 (6) | 1 (1) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/67/NCT04033367/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT04033367/SAP_001.pdf